CLINICAL TRIAL: NCT05989139
Title: Non-Invasive Ventilation And Right Ventricle Function In Cardiogenic Pulmonary Edema: An Echocardiographic Perspective To Select The Appropriate Ventilatory Support
Brief Title: HF vs NIV in Acute Cardiogenic Pulmonary Edema
Acronym: HFvsNIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Sanna Tommaso, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5615
Record Dates: First submitted 2023-06-22; First posted 2023-08-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Edema Cardiac Cause
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPPV (Experimental): non-invasive positive-pressure ventilation arm
  Interventions: Procedure: NPPV/HFNC
- HFNC (Experimental): High-flow nasal cannulae arm
  Interventions: Procedure: HFNC/NPPV

INTERVENTIONS:
Procedure: NPPV/HFNC — Enrolled patients will receive NPPV and HFNC oxygen therapy in a randomized, cross-over fashion, for 40 minutes each. NPPV will be delivered through a full-face mask with a FiO2 starting at 100% and then titrated to achieve an SpO2 of 92-98%. Expiratory positive airway pressure (PEEP) will be firstly set to 5 cmH2O and then increased to a maximum of 15 cmH2O based on SpO2. Pressure support (PS) will be set to an initial value of 10 cmH2O and then increased if signs of respiratory distress persisted or worsened to a maximum value of 20 cmH2O. After 40 minutes, patient is shifted to HFNC ventilation support for 40 minutes.
  At the end of the protocol, the patient will receive the treatment that will be shown as more appropriate for the patient, according to the attending physician, who will be informed about the results of the study on the individual patient.
  Arms: NPPV
Procedure: HFNC/NPPV — Enrolled patients will receive NPPV and HFNC oxygen therapy in a randomized, cross-over fashion, for 40 minutes each.
  HFNC oxygen therapy will start at a flow rate of 60 L/min and will be gradually decreased by 5 cmH2O at time if the patient experienced discomfort. FiO2 will be started at 100% and then titrated to maintain a peripheral oxygen saturation of 92%-98%. Active heating and humidification were provided using MR850, Fisher and Paykel, with a temperature chamber of 37°C. After 40 minutes, patient is shifted to NPPV ventilation support for 40 minutes At the end of the protocol, the patient will receive the treatment that will be shown as more appropriate for the patient, according to the attending physician, who will be informed about the results of the study on the individual patient.
  Arms: HFNC

SUMMARY:
The study's primary aim is

* to compare the effects of two different ventilation modalities, non-invasive positive-pressure ventilation (NPPV) and high-flow nasal cannulae (HFNC), in the acute cardiogenic pulmonary edema (ACPE) setting, in terms of echocardiographic parameters of RV systolic and RV strain.
* to determine the differences of the two interventions on other hemodynamic parameters echocardiographically assessed.
* to assess the differences between the two interventions on physiological parameters, i.e., mean arterial pressure (MAP), heart rate (HR), respiratory rate (RR), oxygen saturation (SpO2), and on arterial blood gases (ABG) analysis parameters (i.e. relief of dyspnea and respiratory distress, patient comfort).

Enrolled patients will receive NPPV and HFNC oxygen therapy in a randomized, cross-over fashion, for 40 minutes each (time 0, T0 and time 1, T1), followed by clinical and echocardiographic evaluation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y.o.;
* Clinical diagnosis of ACPE in the setting of either AMI, acute myocarditis, acute/chronic severe mitral/aortic valve regurgitation, severe mitral/aortic stenosis, acute/chronic HF with rLVEF diagnosed according to European Society of Cardiology (ESC) guidelines [4];
* Hypertensive crisis with systolic blood pressure >200 mmHg;
* Other congenital or acquired structural heart disease causing post capillary pulmonary hypertension or combination of the previous.
* Written informed consent.

Exclusion Criteria:

* Age <18 y.o.;
* Hypercapnia with respiratory acidosis (PaCO2 > 45 mmHg with pH < 7.35);
* History of fever in the previous 4 days;
* White blood cell count > 12.000;
* Increased procalcitonin serum levels;
* Consolidative areas at chest radiograph;
* Hypotension (systolic blood pressure < 85 mmHg);
* Cardiogenic shock;
* Right ventricular (RV) dysfunction;
* Previous cardiac surgery,
* Glasgow Coma Scale score ≤ 8 points;
* Impaired ability to protect the airway from aspiration;
* Orotracheal intubation needed due to cardiopulmonary resuscitation maneuvers;
* Respiratory arrest;
* Severe hemodynamic instability;
* Facial trauma, burns, recent facial surgery or facial anatomy which prevents from the application of the NPPV interface to patient's face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
RV systolic function: Tricuspid annular plane systolic excursion (TAPSE), mm | T0 (Patient's enrollment time)
  Tricuspid annular plane systolic excursion (TAPSE) is a parameter of global RV function which describes apex-to-base shortening. Normal value > 16 mm.
RV systolic function: Tricuspid annular plane systolic excursion (TAPSE), mm | T1 (40 minutes after the first intervention has started)
  Tricuspid annular plane systolic excursion (TAPSE) is a parameter of global RV function which describes apex-to-base shortening. Normal value > 16 mm.
RV systolic function: Tricuspid annular plane systolic excursion (TAPSE), mm | T2 (40 minutes after the second intervention has started)
  Tricuspid annular plane systolic excursion (TAPSE) is a parameter of global RV function which describes apex-to-base shortening. Normal value > 16 mm.
RV systolic function: RV fractional area change (RVFAC), % | T0 (Patient's enrollment time)
  RV fractional area change (RVFAC) is a parameter of radial RV function. It is calculated, in apical four chambers view, as the difference between end-diastolic and end-systolic RV area divided by the end-diastolic area and multiplied by 100. Normal value > 35%.
RV systolic function: RV fractional area change (RVFAC), % | T1 (40 minutes after the first intervention has started)
  RV fractional area change (RVFAC) is a parameter of radial RV function. It is calculated, in apical four chambers view, as the difference between end-diastolic and end-systolic RV area divided by the end-diastolic area and multiplied by 100. Normal value > 35%.
RV systolic function: RV fractional area change (RVFAC), % | T2 (40 minutes after the second intervention has started)
  RV fractional area change (RVFAC) is a parameter of radial RV function. It is calculated, in apical four chambers view, as the difference between end-diastolic and end-systolic RV area divided by the end-diastolic area and multiplied by 100. Normal value > 35%.
RV systolic function: RV Global Longitudinal strain (GLS), % | T0 (Patient's enrollment time)
  RV Global Longitudinal strain (GLS) is an index of systolic performance of RV function. It evaluates the degree of myocardial deformation compared with its original length [L0] (%).
RV systolic function: RV Global Longitudinal strain (GLS), % | T1 (40 minutes after the first intervention has started)
  RV Global Longitudinal strain (GLS) is an index of systolic performance of RV function. It evaluates the degree of myocardial deformation compared with its original length [L0] (%).
RV systolic function: RV Global Longitudinal strain (GLS), % | T2 (40 minutes after the second intervention has started)
  RV Global Longitudinal strain (GLS) is an index of systolic performance of RV function. It evaluates the degree of myocardial deformation compared with its original length [L0] (%).

SECONDARY OUTCOMES:
LV systolic function: Left Ventricle Ejection Fraction (LV EF), % | T0 (Patient's enrollment time)
  Parameter of LV systolic function Normal value > 50%
LV systolic function: Left Ventricle Ejection Fraction (LV EF), % | T1 (40 minutes after the first intervention has started)
  Parameter of LV systolic function Normal value > 50%
LV systolic function: Left Ventricle Ejection Fraction (LV EF), % | T2 (40 minutes after the second intervention has started)
  Parameter of LV systolic function Normal value > 50%
LV diastolic function parameter, i.e. LV average E/E' ratio | T0 (Patient's enrollment time)
  Parameter able to assess LV diastolic function. E/E' ratio normal value < 12.
LV diastolic function parameter, i.e. LV average E/E' ratio | T1 (40 minutes after the first intervention has started)
  Parameter able to assess LV diastolic function. E/E' ratio normal value < 12.
LV diastolic function parameter, i.e. LV average E/E' ratio | T2 (40 minutes after the second intervention has started)
  Parameter able to assess LV diastolic function. E/E' ratio normal value < 12.
Inferior vena cava respiratory variations | T0 (Patient's enrollment time)
  Echocardiographic parameter able to assess fluid responsiveness. Normal value >50%.
Inferior vena cava respiratory variations | T1 (40 minutes after the first intervention has started)
  Echocardiographic parameter able to assess fluid responsiveness. Normal value >50%.
Inferior vena cava respiratory variations | T2 (40 minutes after the second intervention has started)
  Echocardiographic parameter able to assess fluid responsiveness. Normal value >50%.
Physiological parameter: mean arterial pressure (MAP), mmHg | T0 (Patient's enrollment time)
  Normal value >65 mmHg
Physiological parameter: mean arterial pressure (MAP), mmHg | T1 (40 minutes after the first intervention has started)
  Normal value >65 mmHg
Physiological parameter: mean arterial pressure (MAP), mmHg | T2 (40 minutes after the second intervention has started)
  Normal value >65 mmHg
Physiological parameter: oxygen saturation (SpO2), % | T0 (Patient's enrollment time)
  Normal value > 90%
Physiological parameter: oxygen saturation (SpO2), % | T1 (40 minutes after the first intervention has started)
  Normal value > 90%
Physiological parameter: oxygen saturation (SpO2), % | T2 (40 minutes after the second intervention has started)
  Normal value > 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico Agostino Gemelli Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No